CLINICAL TRIAL: NCT02975908
Title: A Realworld Study of Acute Respiratory Distress Syndrome in China
Acronym: CHARDSnet
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: PLA General Hospital (Unknown); Second Xiangya Hospital of Central South University (Other); Xiangya No.1 Hospital of Central South University (Unknown); The Second Affiliated Hospital of Chongqing Medical University (Other); Beijing Chao Yang Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Hospital Affiliated to China Medical University (Unknown); Nanjing General Hospital (Unknown); Peking University First Hospital (Other); Third Hospital Affiliated to Neimenggu Medical University (Unknown); Second Hospital Affiliated to Hebei Medical University (Unknown); Qilu Hospital of Shandong University (Other); First Hospital Affiliated to Anhui Medical University (Unknown); Ruijin Hospital (Other); Beijing Hospital (Other Government); Peking Union Medical College Hospital (Other); No.3 Hospital of Peking University (Unknown); Fuxing Hospital (Unknown); Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Chen Wang, professor, China-Japan Friendship Hospital
Other Study IDs: CHARDS20160301
Record Dates: First submitted 2016-04-05; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; epidemiology; clinical features; management; prognosis
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
ARDS is a critical respiratory disease caused by endogenous and exogenous factors. The mortality of ARDS varies from 30 to 70%. In 2012, a new international diagnostic criterion has been put forward. Yet, its feasibility, reliability and validity need to be tested. Meanwhile, the correlation of different severity and prognosis remains unclear. As so far, the epidemiological information about ARDS in China is lacking.

Investigators plan to conduct a multi-center observational study（real-life study） to investigate the risk factors, morbidity, management and prognosis of ARDS in China, in order to facilitate standardization of diagnosis and management of ARDS and provide basic data and idea for further clinical intervention studies.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age; hospitalized patients with main diagnosis as ARDS.

Exclusion Criteria:

* <18 years of age
* Patients or their families refused to participate in the study
* Patients diagnosed as COPD, pulmonary fibrosis or bronchiectasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research plans to enroll 400 hospitalized patients (≥ 18 years old with main diagnosis as ARDS). Sample size estimation is based on estimated mortality of ARDS hospitalized patients (~5%). Study patients will be recruited from 20 hospitals across China,each hospital will recruit 20 patients. Hospital selection follows a multi-stage sampling strategy.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28days
  the 28days mortality after the diagnosis of ARDS

SECONDARY OUTCOMES:
Length of ICU stay | 90 days
  The days between admission to intensive care unit(ICU) and discharge from ICU.
Ventilation free days | 28 days
  The days between successful weaning from mechanical ventilation and day 28 after study enrollment.
Incidence of ARDS | 2 years
  The total number of acute respiratory distress syndrome(ARDS)patients in 2 years.
Severity of patients | 2 years
  Number of patients in each grade of severities according to Berlin definition: the number of mild, moderate and severe acute respiratory distress syndrome(ARDS) patients will be recorded.
Adverse events related to treatment | 90 days
  Number of patients with adverse events, include biotrauma, worsen of hemodynamics, hospital-acquired infection, patient-ventilator asynchrony, gastric distention, aspiration etc.
Number of patients using adjuvant drugs | 28 days
  Adjuvant drugs refer to corticosteroid, sedative, analgesic and non depolarizing muscle relaxant.
Number of patients with high risk factors | 1 week
  High risk factors for acute respiratory distress syndrome(ARDS), including endogenous factors as pneumonia, aspiration, lung contusion and drowning; the exogenous factors as extrapulmonary trauma, extra pulmonary sepsis , hypovolemic shock, pancreatitis, severe burning, drug overdose, blood transfusion，eclampsia etc.
Number of patients with conventional respiratory support techniques | 28 days
  Conventional respiratory support techniques include noninvasive positive pressure ventilation(NPPV), invasive positive pressure ventilation(include volume-controlled ventilation and pressure-controlled ventilation) .
Number of patients with unconventional respiratory support techniques | 28 days
  Unconventional respiratory support techniques include recruitment maneuver(RM), prone position ventilation(PPV), high-frequency oscillatory ventilation(HFOV) ,extracorporeal membrane oxygenation(ECMO) and extracorporeal CO2 removal(ECCO2R)
Number of patients with impaired lung function | 90 days, 1 year
  The number patients with impaired lung function 90 days and 1 year after diagnosis of acute respiratory distress syndrome(ARDS).
Number of patients with abnormal lung CT | 90 days, 1 year
  The number patients with abnormal lung CT 90 days and 1 year after diagnosis of acute respiratory distress syndrome(ARDS).

CONTACTS AND LOCATIONS:
Locations (1):
- China - Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang H, Xia J, Huang X, Bai Y, Jin D, Nouraie SM, McVerry BJ, Morris A, Kitsios GD, Wang C, Zhan Q. Generalisability of ARDS biological subphenotype models in Asians: an international, multicentre, prospective biomarker study. Thorax. 2025 Oct 29:thorax-2025-223421. doi: 10.1136/thorax-2025-223421. Online ahead of print. PMID 41167619
- [Derived] Huang X, Zhang R, Fan G, Wu D, Lu H, Wang D, Deng W, Sun T, Xing L, Liu S, Wang S, Cai Y, Tian Y, Zhang Y, Xia J, Zhan Q; CHARDSnet group. Incidence and outcomes of acute respiratory distress syndrome in intensive care units of mainland China: a multicentre prospective longitudinal study. Crit Care. 2020 Aug 20;24(1):515. doi: 10.1186/s13054-020-03112-0. PMID 32819400